CLINICAL TRIAL: NCT01494350
Title: Open-label Treatment of Non-complicated, Non-severe, Cutaneous Leishmaniasis in Tunisia With WR 279,396 (Paromomycin + Gentamicin Topical Cream) )
Brief Title: WR 279,396 Open Label Treatment Protocol in Tunisia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed prematurely due study team travel restrictions.
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-10-0006; A-16898.3
Record Dates: First submitted 2011-11-30; First posted 2011-12-19 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous leishmaniasis; topical treatment; Tunisia
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WR 279,396 topical cream (Experimental): 120 subjects will be enrolled to this open label study to receive WR 279,396 topical cream
  Interventions: Drug: WR 279,396 topical cream

INTERVENTIONS:
Drug: WR 279,396 topical cream — WR 279,396 is a topical antibiotic cream containing paromomycin and gentamicin that will be applied to each lesion once a day for 20 days and covered with a sterile gauze and tape dressing.
  Other Names: WR 279, 396; Topical Paromomycin + Gentamicin Cream

SUMMARY:
The U.S. Army has recently completed a Phase 3 clinical trial in Tunisia. This is an open-label single site trial designed to expand our safety database and capture additional efficacy (final clinical cure rate of an index lesion) of WR 279,396 Topical Cream in Tunisian subjects with non-complicated, non-severe Cutaneous Leishmaniasis (CL). Subjects will be patients who visit Ministry of Health sponsored clinics in Tunisia who present with at least one CL lesion that is ulcerated and amenable to topical treatment. Potential trial subjects will be consented and screened for eligibility including medical history, physical exam, lesion parasitology, and renal and liver function tests. If eligible for the study, subjects will receive WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) (target n = 110). The cream will be applied topically to all CL lesions once daily for 20 days by an investigator or study nurse. If a subject develops a new lesion during the study, the new lesion may also be treated with the topical cream.

DETAILED DESCRIPTION:
Subjects will have an in-clinic follow-up on Days 28 +/- 2 days, 42 +/- 4 days and 98 +/- 8 days to assess safety and cure rates. Safety variables including adverse events (AEs) and serious adverse events (SAEs) will be collected through Day 98. For the primary efficacy evaluation, the index ulcerative lesion will be assessed for clinical response by measurement of the length and width of area of ulceration. All other treated lesions will also be assessed for cure as secondary efficacy endpoints with ulcerated and non-ulcerated lesions being evaluated independently. An ulcerated lesion will be considered to be completely cured if 100% reepithelialization is observed. The length and width of non-ulcerated lesions (nodules, plaques) will also be measured and evaluated for cure (ie, absence of signs of an active lesion). The primary efficacy endpoint is the final clinical cure rate calculated by the number of index lesions that had 100% reepithelialization at Day 98 divided by the total number of index lesions that received at least one topical treatment of WR 279,396.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Subject has a diagnosis of CL in at least one lesion by at least one of the following methods: 1) microscopic identification of amastigotes in stained lesion tissue, or 2) positive culture for promastigotes.
* Subject has a parasitologically confirmed lesion that satisfies the following criteria for an Index lesion:

  * ulcerative in character
  * lesion size ≥ 1 cm and ≤5 cm (including the area of induration surrounding the lesion)
  * not located on the ear, or on a location that in the opinion of the PI is difficult to maintain application of study drug topically.
* Subject has < 7 leishmaniasis total lesions.
* Subject is willing to forego other forms of treatments for CL including other investigational treatments during the study.
* In the opinion of the investigator, the subject (or their legal guardian) is capable of understanding and complying with the protocol.

Exclusion Criteria:

* Female with a positive serum pregnancy test or who is breast feeding.
* History of clinically significant medical problems in the investigator's judgment that might interact, either negatively or positively, with topical treatment of leishmaniasis including any immunocompromising condition.
* Age adjusted blood creatinine or blood urea nitrogen (BUN) levels indicative of clinically significant renal disease or aspartate amino transferase (AST), alanine amino transferase (ALT), or total bilirubin that suggest clinically significant hepatic impairment as judged by the PI or subinvestigator. Note: This study is designed to evaluate populations who may have some renal or hepatic dysfunction as the drug has not been shown to have serum levels that would be expected to show renal or hepatic toxicity and treatment of the general population presenting with CL is highly desired based on its safety profile compared to other leishmanial drugs.
* Evidence of disseminated leishmaniasis.
* Received treatment for leishmaniasis with antimonials or any medication likely, in the opinion of the PI, to modify the course of the Leishmania infection within 56 days of starting study treatments.
* History of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afif Ben Salah, M.D., Ph.D., Principal Investigator — Institute Pasteur Tunisia
Locations (1):
- Central Clinic-Sidi Bouzid, Tunis, Tunisia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 184 total screened and there were 134 screen failures.
Period: Overall Study
Arm/Group | WR 279,396 Topical Cream
Started | 50
Completed | 49
Not Completed | 1
Not completed — Worsening of lesion | 1

BASELINE CHARACTERISTICS:
Population: modified intent to treat (mITT)/safety subjects
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  North African | 50
Number of lesions per subject [Mean (Standard Deviation); unit: lesions] | 1.96 (1.48)

OUTCOME MEASURES:

1. Primary Outcome: Final Clinical Cure Rate for the Index Lesion
Description: Number of index lesions with 100% reepithelialization at Day 98.
Time Frame: Final clincial cure is measured at day 98
Population: modified intent to treat (mITT)
Measure: Number; unit: lesions
Units Other Than Participants: index lesions
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 50
Number analyzed (index lesions) | 50
lesions | 48

2. Secondary Outcome: Area of Index Lesions Throughout the Study
Description: Area (mm^2) of index lesion on Days 0, 20, 28, 42, and 98.
Time Frame: Measured at day 0, 20, 28, 42, and 98
Population: modified intent to treat (mITT). Baseline for this outcome measure does not include one subject (1 index lesion) who withdrew on Day 18.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Index lesions
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 49
Number analyzed (Index lesions) | 49
mm^2
  Baseline (Day 0) | 121 (106)
  Day 20 | 393 (315)
  Day 28 | 203 (238)
  Day 42 | 38.9 (83.2)
  Day 98 | 7.88 (55.1)

3. Secondary Outcome: Number of Index Lesions With Reepithelialization Throughout the Study
Description: Number of index lesions with 100% reepithelialization on Days 28 and 42.
Time Frame: Measured at day 28 and 42
Population: modified intent to treat (mITT). This outcome measure does not include one subject (2 lesions) who withdrew on Day 18.
Measure: Number; unit: lesions
Units Other Than Participants: Index lesions
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 49
Number analyzed (Index lesions) | 49
lesions
  Day 28 | 8
  Day 42 | 28

4. Secondary Outcome: Area of All Ulcerated Lesions Throughout the Study
Description: Area of all ulcerated lesions on Days 20, 28, 42, and 98.
Time Frame: Measured at day 20, 28, 42 and 98
Population: modified intent to treat (mITT). Baseline for this outcome measure does not include one subject (2 lesions) who withdrew on Day 18.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: lesions
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 49
Number analyzed (lesions) | 96
mm^2
  Baseline (Day 0) | 82.6 (90.4)
  Day 20 | 288 (275)
  Day 28 | 149 (198)
  Day 42 | 22.1 (63.3)
  Day 98 | 4.02 (39.4)

5. Secondary Outcome: Number of All Ulcerated Lesions With Reepithelialization on Day 28
Description: Final cure rate for all ulcerated lesions (100% reepithelialization for ulcerative lesions) on Day 28
Time Frame: Measured on day 28
Population: modified intent to treat (mITT). This outcome measure does not include one subject (2 lesions) who withdrew on Day 18.
Measure: Number; unit: lesions
Units Other Than Participants: Lesions
Arm/Group | WR 279,396 Topical Cream
Number analyzed (Participants) | 49
Number analyzed (Lesions) | 96
lesions | 23

ADVERSE EVENTS:
Time Frame: 98 days
Arm/Group | WR 279,396 Topical Cream
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 39/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WR 279,396 Topical Cream (N=50)
Application site erythema (General disorders) | 12
Application site vesicles (General disorders) | 27
Oedema (General disorders) | 1
Pain (General disorders) | 1
Bronchitis acute (Infections and infestations) | 2
Superinfection (General disorders) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotrasnsferase increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 10
Skin irritation (Skin and subcutaneous tissue disorders) | 9

LIMITATIONS AND CAVEATS:
This study was closed prematurely due study team and travel restrictions but not due to any safety issues with the study subjects. Only a total of 50 of the 110 planned subjects were enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No